CLINICAL TRIAL: NCT05253794
Title: Effect of Colchicine on the Progression of Aortic Valve Stenosis - a Pilot Study
Acronym: COPAS-Pilot
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20210526
Record Dates: First submitted 2022-02-01; First posted 2022-02-24 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Aortic Stenosis; Inflammation
Keywords: colchicine
MeSH Terms: conditions — Aortic Valve Stenosis; Inflammation | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Experimental): Colchicine 0.6mg PO daily for 6 months
  Interventions: Drug: Colchicine 0.6 mg
- Placebo (Placebo Comparator): Placebo tablet daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine 0.6 mg — oral tablet daily for 6 months
  Arms: Colchicine
Drug: Placebo — oral tablet daily for 6 months
  Arms: Placebo

SUMMARY:
COPAS pilot is a pilot single center double blinded randomized study to determine the effect of targeted anti-inflammation therapy using colchicine, on valvular calcification activity using imaging, i.e. aortic valvular NaF uptake. The current proposal uses a randomized design to evaluate the effect of colchicine vs. placebo on valvular calcification activity over 6 months measured using NaF PET

DETAILED DESCRIPTION:
COPAS pilot is a pilot single center double blinded randomized study. The investigators will compare the effect of colchicine (0.6 mg daily - intervention arm) vs. placebo (control group) on the 18F NaF aortic valve uptake in patients with mild to moderate AS defined by a mean pressure gradient measured using transthoracic echocardiography (TTE) between 15-25 mm Hg after a 6-month period of treatment. The investigators plan to enroll 12 patients (6 males/6 females) in each arm (total sample size: 24 patients). Primary endpoint is the change in 18FNaF aortic valve uptake between baseline and 6 months in each arm. Parameters of interest are the maximal and total standard uptake values (SUVs) and tissue-to background ratios (TBRs) at the level of the aortic valve.

ELIGIBILITY:
Inclusion Criteria:

1. mild to moderate aortic stenosis defined by a mean pressure gradient using transthoracic echocardiography (TTE) between 15-25mmHg.
2. age greater than18 years;
3. given informed consent.

Exclusion Criteria:

1. bicuspid aortic valve
2. associated moderate to severe aortic regurgitation
3. associated other valvular pathology of moderate or greater severity
4. LV dysfunction (EF<50%);
5. decompensated heart failure;
6. active infection (e.g. pneumonia, active skin infections, and on antibiotics);
7. chronic diarrhea;
8. immune compromise (e.g. recurrent infection);
9. history of cancer within the last 3 years (other than a successfully treated cutaneous squamous cell or basal cell carcinoma or localized carcinoma in situ of the cervix).
10. active inflammatory conditions (e.g. rheumatoid arthritis, chronic inflammatory bowel disease, SLE, systemic anti-inflammatory therapy (e.g. prednisone, methotrexate));
11. pregnancy (all women of child bearing potential will have a negative BHCG test;
12. breastfeeding;
13. Women of childbearing potential who refuse to use two forms of contraception (this includes at least one form of highly effective and one effective method of contraception) throughout the study OR men capable of fathering a child who refuse to use contraception.
14. glomerular filtration rate (GFR) <50 ml/min/1.72m2;
15. Use of p-glycoprotein inhibitor (e.g. cyclosporine, verapamil, or quinidine) or a strong CYP3A4 inhibitor (e.g. ritonavir, clarithromycin, or ketoconazole);
16. Hemoglobin < 105(women) <110 (men) g/L; WBC < 3.0x 10(9)/L, platelet count< 110x 10(9)/L;
17. Patient with a history of cirrhosis, chronic active hepatitis or severe hepatic disease or with alanine aminotransferase (ALT) levels greater than 3 times the upper limit of normal.
18. unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in aortic valve calcification activity | 6 months
  Change in valvular calcification activity as measured by NaF uptake by Target to Background Ratio (TBR) on PET/CT imaging

OTHER OUTCOMES:
Change in aortic valve calcification | One year
  Change is the degree of aortic valve calcification measured using CT scan (calcium score) and expressed in arbitrary units

CONTACTS AND LOCATIONS:
Overall Officials: David Messika-Zetioun@ottawaheart.ca, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No